CLINICAL TRIAL: NCT06870708
Title: Arthroscopic Repair Of Partial Thickness Articular Side Rotator Cuff Tears Using Transtendon Versus Conversion Repair Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed hussein khalil, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-383-2023
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Tears
Keywords: Partial thickness rotator cuff tear; Transtendon technique; conversion technique.
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: prospective comparative study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Conversion repair technique: Group A (Experimental): arthroscopic repair of partial rotator cuff tear using the conversion technique
  Interventions: Procedure: arthroscopic repair of partial rotator cuff tear using the conversion versus the transtendon technique
- The Transtendon repair technique: Group B (Experimental): arthroscopic repair of partial rotator cuff tear using the transtendon technique
  Interventions: Procedure: arthroscopic repair of partial rotator cuff tear using the conversion versus the transtendon technique

INTERVENTIONS:
Procedure: arthroscopic repair of partial rotator cuff tear using the conversion versus the transtendon technique — arthroscopic repair of partial rotator cuff tear using the conversion versus the transtendon technique

SUMMARY:
This study aims to compare the functional results of patients who underwent two different arthroscopic methods for the management of articular-sided partial-thickness rotator cuff tears (PT-RCTs).

The present study aims to compare the functional results following the repair of PT-RCTs using the conversion versus the trastendon techniques

DETAILED DESCRIPTION:
This is a prospective randomized study carried out at a tertiary trauma center between October 2022 and June 2023. The research ethical Committee authorized this study protocol [(Institutional Review Board (IRB) number: N-383-2023)], and all participants signed an informed consent prior to joining the study. This study included 50 patients with PT-RCTs who underwent arthroscopic repair using either the conversion technique (25 patients) in group A or the transtendon technique (25 patients) in group B. The random assignment of all patients to enter either group was computerized using simple randomization.

ELIGIBILITY:
The inclusion criteria were:

* Patients suffering symptomatic PT-RCTs exceeding 50% of the tendon thickness, documented by preoperative magnetic resonance imaging (MRI) and confirmed by arthroscopy intraoperative.
* Failure of nonoperative management for at least 3 months.

The exclusion criteria were:

* Prior shoulder surgery.
* Severe concomitant pathologies including glenohumeral arthritis, advanced subscapularis tear, and biceps tendon rupture.
* Associated Bankart lesion.
* Patients with uncontrolled Diabetes mellites.

Ages: 49 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons score | baseline, and 18 months after surgery
  shoulder score, the maximum is 100, the minimum is zero, a higher score means a better outcome
Constant and Murley score | baseline, and 18 months after surgery
  shoulder score, the maximum is 100, the minimum is zero, a higher score means a better outcome

SECONDARY OUTCOMES:
Visual analogue scale | baseline, and 18 months after surgery
  pain score, the minimum is zero, the maximum is 10, the higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H khalil, M.D, Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang Y, Hu D, Chen S, Guan S, Shang X. Transtendon technique versus repair after completion of the tear for articular-sided partial rotator cuff tear: a meta-analysis of comparative studies. J Orthop Surg Res. 2023 May 22;18(1):378. doi: 10.1186/s13018-023-03831-4. PMID 37217901
- [Background] Thamrongskulsiri N, Limskul D, Itthipanichpong T, Tanpowpong T, Kuptniratsaikul S. Similar outcomes between transtendon repair and tear completion repair techniques for partial articular-sided supraspinatus tendon avulsion lesions: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2023 Oct;31(10):4575-4584. doi: 10.1007/s00167-023-07502-z. Epub 2023 Jul 15. PMID 37452830
- [Background] Sun L, Zhang Q, Ge H, Sun Y, Cheng B. Which is the best repair of articular-sided rotator cuff tears: a meta-analysis. J Orthop Surg Res. 2015 May 28;10:84. doi: 10.1186/s13018-015-0224-6. PMID 26016477
- [Background] Shin SJ. A comparison of 2 repair techniques for partial-thickness articular-sided rotator cuff tears. Arthroscopy. 2012 Jan;28(1):25-33. doi: 10.1016/j.arthro.2011.07.005. Epub 2011 Oct 14. PMID 22000411
- [Background] Castagna A, Borroni M, Garofalo R, Rose GD, Cesari E, Padua R, Conti M, Gumina S. Deep partial rotator cuff tear: transtendon repair or tear completion and repair? A randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):460-3. doi: 10.1007/s00167-013-2536-6. Epub 2013 May 21. PMID 23689964